CLINICAL TRIAL: NCT00576589
Title: A Phase 1, 2-Part, Randomized, Subject And Investigator Blinded, Placebo-Controlled, Cross-Over Trial To Evaluate The Safety, Tolerability And Pharmacokinetics Of CE-326,597 In Obese, Adult Subjects With Asymptomatic Cholelithiasis
Brief Title: Study Of The Safety And Pharmacokinetics Of CE-326,597 In Patients With Asymptomatic Gallstones
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7211006
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2008-11

CONDITIONS: Obesity
Keywords: Safety in patients with Asymptomatic cholelithiasis/gallstones.
MeSH Terms: conditions — Obesity; Gallstones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CE-326,597 (Experimental)
  Interventions: Drug: CE-326,597
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CE-326,597 — CE-326,597 administered orally, once daily for 14-days at 1 to 2 doses (25 mg QD, 100 mg QD) with the morning meal.
  Arms: CE-326,597
Drug: Placebo — CE-326,597 matching placebo administered orally, once daily for 14-days with the morning meal.
  Arms: Placebo

SUMMARY:
The study is designed to assess whether repeated dosing with CE-326,597 will cause patients with asymptomatic gallstones (as detected on screening abdominal ultrasound) to become symptomatic. In addition, the study will characterize the pharmacokinetics of CE-326,597.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 30-40 kg/m2, inclusive
* Evidence of asymptomatic cholelithiasis on screening abdominal ultrasound

Exclusion Criteria:

* Patients with unstable medical conditions, such as diabetes, stroke, heart attack.
* Females of childbearing potential or those who may be pregnant or breast feeding.
* Patients with inflammed gallbladder, evidence of stones in bile ducts on screening abdominal ultrasound, history of symptoms indicating active gallbladder disease or gallbladder removal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed via AEs/SAEs, plus where applicable gastrointestinal symptoms checklist, clinical laboratory tests, vital signs (blood pressure and pulse rate) | Day 1 to 14
CE-326,597 pharmacokinetics by estimating AUC0-24, Cmax and Tmax | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Willingboro, New Jersey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7211006&StudyName=Study%20Of%20The%20Safety%20And%20Pharmacokinetics%20Of%20CE-326%2C597%20In%20Patients%20With%20Asymptomatic%20Gallstones